CLINICAL TRIAL: NCT06135623
Title: Long-Term Impact of COVID-19 Restrictions on Physical Activity and Social Interactions in Young Adults
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Gökhan Can TÖRPÜ, Principal Investigator, Bezmialem Vakif University
Other Study IDs: BezmialemVU-GCT-03
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: COVID-19; Social Interaction; Physical Inactivity
Keywords: COVID-19 restrictions; Physical activity; Social interactions; Young adults
MeSH Terms: conditions — COVID-19; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 Group: Having a history of COVID-19 infection
- Non-COVID-19 Group: No history of COVID-19 infection

SUMMARY:
There are studies on the impact of quarantine measures taken during the COVID-19 pandemic on individuals' social interactions and physical activities. We think that the adaptation of individuals who have had COVID-19 infection to return to social and physical activities after restrictions may affect participation in these activities. The aim of this study is to investigate the long-term impact of COVID-19 restrictions on physical activity and social interaction in young adults, depending on whether they have had a COVID-19 infection.

DETAILED DESCRIPTION:
Corona Virus Disease-19 was declared as a pandemic on 11 March 2020 by the World Health Organization. The fact that the measures taken to prevent the spread of the pandemic bring about a global quarantine process affects people's social interactions and physical activity levels with each other. The aim of this study is to investigate the long-term impact of COVID-19 restrictions on physical activity and social interaction in young adults, depending on whether they have had a COVID-19 infection. Physical activity levels were assessed with the short form of the International Physical Activity Questionnaire-Short Form. Social interactions and social phobias are Social Interaction Anxiety Scale and Social Phobia Scale were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Young adults aged 18-25
* Agreeing to participate in the study

Exclusion Criteria:

* Having mental retardation

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young adults aged 18-25
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Social Interaction Anxiety Scale (SIAS) | Four Months
  The social interaction anxiety level of the participants was measured with the Social Interaction Anxiety Scale (SIAS).
Social Phobia Scale (SPS) | Four Months
  Social phobia levels of the participants were evaluated using the Social Phobia Scale (SPS)
International Physical Activity Questionnaire Short Form | Four Months
  The short form of the International Physical Activity Questionnaire (IPAQ-SF) was used to determine the physical activity levels of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan C Törpü, BPT, Study Chair — Bezmialem Vakif University; Müberra Tanrıverdi, PhD, Study Director — Bezmialem Vakif University; Nahide Öztoprak, BPT, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Eyüp, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mattick RP, Clarke JC. Development and validation of measures of social phobia scrutiny fear and social interaction anxiety. Behav Res Ther. 1998 Apr;36(4):455-70. doi: 10.1016/s0005-7967(97)10031-6. PMID 9670605
- [Background] Saglam M, Arikan H, Savci S, Inal-Ince D, Bosnak-Guclu M, Karabulut E, Tokgozoglu L. International physical activity questionnaire: reliability and validity of the Turkish version. Percept Mot Skills. 2010 Aug;111(1):278-84. doi: 10.2466/06.08.PMS.111.4.278-284. PMID 21058606
- [Background] Woods JA, Hutchinson NT, Powers SK, Roberts WO, Gomez-Cabrera MC, Radak Z, Berkes I, Boros A, Boldogh I, Leeuwenburgh C, Coelho-Junior HJ, Marzetti E, Cheng Y, Liu J, Durstine JL, Sun J, Ji LL. The COVID-19 pandemic and physical activity. Sports Med Health Sci. 2020 Jun;2(2):55-64. doi: 10.1016/j.smhs.2020.05.006. Epub 2020 May 30. PMID 34189484